CLINICAL TRIAL: NCT01578928
Title: A Phase I, Open-label, Multicenter, Single Dose Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous (s.c.) Pasireotide in Subjects With Varying Degrees of Renal Impairment Compared to a Matched Control Group of Healthy Volunteers
Brief Title: A Phase l Study to Evaluate the Pharmacokinetics and Safety Pasireotide in Subjects With Varying Degrees of Renal Impairment Compared to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2126; 2011-005922-23 (EudraCT Number)
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-09

CONDITIONS: Renal Impairment
Keywords: renal, impairment, endstage renal disease; renal; impairment; endstage renal disease
MeSH Terms: conditions — Renal Insufficiency | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOM230 (Experimental): subjects with varying degrees of renal impairment along with subjects without renal impairment
  Interventions: Drug: SOM230

INTERVENTIONS:
Drug: SOM230

SUMMARY:
The purpose of this study is to assess the effect of renal impairment on the pharmacokinetics (PK) of pasireotide,the PK of pasireotide in subjects with different degrees of renal impairment.

DETAILED DESCRIPTION:
This is a phase I, open-label, multicenter, single dose study to evaluate the PK and safety of pasireotide s.c. injection in subjects with varying degrees of renal impairment compared to healthy subjects with normal renal function. Subjects will be classified by their respective degree of renal functions (normal, mild, moderate, severe, and ESRD (End Stage Renal Disease) according to eGFR as determined at the screening visit.

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for inclusion in this study have to meet all of the following criteria:

1. Written informed consent obtained prior to any screening procedures.
2. Subjects must be able to communicate well with the investigator and comply with the requirements of the study procedures
3. Male or female subjects between 18 and 75 years of age, inclusive.
4. Vital Signs at screening and baseline which are within the following ranges:

   * Oral body temperature: ≥ 35.0 and ≤ 37.5 ˚C
   * Pulse rate: 40-90 bpm
5. Subjects must have a BMI between 20 kg/m2 and 30 kg/m2 and weigh at least 50 kg and no more than 120 kg.
6. Subjects must be willing to comply with dietary, fluid, and lifestyle restrictions (from day-1 to study completion).
7. Other than renal impairment, subjects must be stable and appropriately managed relative to chronic diseases (such as diabetes and hypertension) as determined by past medical history, physical examination, electrocardiogram, and laboratory tests for chemistry and hematology.

   For renal impairment subjects only
8. Subjects must have stable renal disease without evidence of renal progressive disease (stable renal disease is defined as no significant change, such as, stable eGFR, for 12 weeks prior to study entry).
9. Blood pressure (3 minutes resting before measurement) in the supine position:

   * Systolic: 90-165 mmHg
   * Diastolic: 60-110 mmHg

   For control subjects only
10. Subjects must be matched to at least one renal impaired subject by gender, age (±10 years), body weight (±20%), BMI (±5%) and race.
11. Blood pressure (3 minutes resting before measurement) in the supine position:

    * Systolic: 90-140 mmHg
    * Diastolic: 50-90 mmHg

Exclusion criteria:

Subjects eligible for this study must not meet any of the following criteria:

1. Clinically significant abnormal laboratory values at the screening evaluation or at the baseline re-evaluation, excluding those normally associated with mild to severe degree of renal impairment or the primary cause of renal insufficiency
2. Use of any over-the-counter medications or vitamins or herbal/natural supplements during 2 weeks prior to dosing (acetaminophen is acceptable, and must be documented in the Concomitant Medications/Non-Drug Therapies page of the CRF)
3. Current medical history of the following:

   * Sustained or clinically significant cardiac arrhythmias
   * History of syncope or family history of idiopathic sudden death
   * Risk factors for torsades de pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high grade AV block
   * Screening QTcF > 450ms
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * Concomitant medications known to increase the QT interval
4. Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation
5. Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing or other amount considered to compromise the health of the subject if previous history of anemia exists
6. Significant acute illness within the two weeks prior to dosing
7. History of immunocompromise, including a positive HIV (ELISA and Western blot) test result
8. History of allergies to the investigational compound/compound class being used in the study
9. A positive Hepatitis B surface antigen (HBsAg) or positive HCV antibody
10. History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations
11. History of liver disease, such as cirrhosis or chronic active hepatitis B and C.
12. Known gallbladder or bile duct disease, acute or chronic pancreatitis
13. Baseline ALT or AST > ULN
14. Baseline total bilirubin > 1.5x ULN
15. Subjects on dialysis
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 5 times the terminal half-life of study treatment (6 days). Highly effective contraception methods include:

    * Total abstinence or
    * Male or female sterilization or
    * Combination of any two of the following (a+b or a+c, or b+c):

      * Use of oral, injected or implanted hormonal methods of contraception
      * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
17. Sexually active males unless they use a condom during intercourse while taking drug and for 5 half-lives (6 days) after stopping SOM230 medication and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
18. Potentially unreliable or vulnerable subjects (e.g. person kept in detention) and those judged by the investigator to be unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Plasma and Urine PK parameters | pre-dose (-1 min) and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10 and 12, 24, 36, 48, 72, 96, 120 and 122 hours post-dose
  Description: Cmax, AUCinf, AUClast, CL/F, CLR, glucose, insulin, glucagon

SECONDARY OUTCOMES:
Additional PK parameters | pre-dose (-1 min) and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 24, 36, 48, 72, 96, 120 and 122 hours post-dose
  Description: Vz/F, T1/2, Fu, Cmax,u, AUCinf,u, AUClast,u, CLu/F and Vu/F

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Bloemfontein, Free State, South Africa

REFERENCES:
- See also: Results for CSOM230B2126 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13770